CLINICAL TRIAL: NCT05621135
Title: Validity and Reliability of the Sitting Assessment Scale in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Demet GÖZAÇAN KARABULUT, Assistant Professor, Gaziantep Islam Science and Technology University
Other Study IDs: GIBTU-FTR-DGK-2
Record Dates: First submitted 2022-11-04; First posted 2022-11-17 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Validity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Sitting Assessment Scale is a valid and reliable scale that evaluates sitting balance in Cerebral Palsy (CP). The validity and reliability study of the scale has been done, but it has not been adapted to Turkish language. The aim of this study is to adapt the Sitting Evaluation Scale, which evaluates sitting balance in Cerebral Palsy, into Turkish and to examine the validity and reliability of the Turkish version of the scale.

DETAILED DESCRIPTION:
Cerebral Palsy will be participate the study between the ages of 2 and 18 years. Children's classified with GMFCS and MACS.

Evaluation will be applied to the volunteer participants after the translation steps of the Sitting Evaluation Assessment are completed. The validity of the scale will be examined in terms of construct validity and content validity. All evaluations will be performed in the clinic with the specialist physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cerebral Palsy voluntary participation,
* Age between 2-18 years

Exclusion Criteria:

* Not voluntary to participate in the research,
* Botox in the last 6 months,
* Hip or spine surgeries in the last 6 months

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cerebral Palsy will be participate the study between the ages of 2 and 18 years.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | At Baseline
  Assessing functional level and motor functions of children with CP.
Manuel ability classification system (MACS) | At Baseline
  This is a classification system based on the grasping and releasing objects in daily life, and how they use their hands while holding objects. It is classify the hand skills of children with CP between the ages of 4-18.Children with CP are classified in five levels with MACS. The higher level indicates worse hand function.
Gross Motor Function Measure-88 | At Baseline
  It is used to show gross motor functions and changes in these functions. It consists of five main sections. Each section can be used by calculating separately within itself. The total score ranges from 0 to 100, with a high score indicating better function.
Trunk Control Measurement Scale | At Baseline
  This scale consists of two main parts as dynamic and static sitting balance. The scale consists of 15 questions. The scoring of the items is 0, 1, 2 or 3. The total score ranges from 0 to 58, with a high score indicating better trunk control.
Sitting Assessment Scale | At Baseline and 2 weeks after the baseline
  The Sitting Assessment Scale is a standard observation tool designed for the assessment of sitting in children with CP. The scale consists of five items evaluating head, trunk and foot control and arm and hand functions.The lowest score that can be obtained from the scale is 5 and the highest score is 20. It can be stated that higher scores better functions.

CONTACTS AND LOCATIONS:
Overall Officials: Demet GÖZAÇAN KARABULUT, Study Director — Gaziantep Islam Science and Technology University
Locations (1):
- Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No